CLINICAL TRIAL: NCT04062890
Title: Inhibiting GABA Transaminase to Relieve Obesity Induced Hyperinsulinemia and Insulin Resistance
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was never opened at University of Arizona.
Sponsor: University of Arizona (Other)
Collaborators: Arizona Department of Health Services (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADHS18-201472b
Record Dates: First submitted 2019-08-15; First posted 2019-08-20 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2024-05

CONDITIONS: Hyperinsulinism; Insulin Resistance; Insulin Sensitivity; Glucose Intolerance; Hypertension
Keywords: Type II Diabetes; Hyperinsulinism; Insulin Resistance; Hypertension
MeSH Terms: conditions — Hyperinsulinism; Insulin Resistance; Glucose Intolerance; Hypertension; Diabetes Mellitus, Type 2 | interventions — Vigabatrin

STUDY DESIGN:
Intervention Model Description: Patients will be treated with a placebo or vigabatrin
Who Masked: Participant, Care Provider, Investigator
Masking Description: Only the pharmacist and the principle investigator will know the treatments designated to a patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vigabatrin (Active Comparator): Vigabatrin - Pill, 500 mg twice daily for 7 days (days 1-7), 1000 mg twice daily for 7 days (days 8-14), 1500 mg twice daily for 10 days (days 15-24), 1000 mg twice daily for 7 days (days 25-31), 500 mg twice daily for 7 days (days 32-38).
  Interventions: Drug: Vigabatrin Pill
- Placebo (Placebo Comparator): Placebo - Pill, 1 pill twice daily for 7 days (days 1-7), 2 pills twice daily for 7 days (days 8-14), 3 pills twice daily for 10 days (days 15-24), 2 pills twice daily for 7 days (days 25-31), 1 pill twice daily for 7 days (days 32-38).
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Vigabatrin Pill — Oral Vigabatrin Pill
  Arms: Vigabatrin
Drug: Placebo oral tablet — Oral Placebo Pill
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
50% of Arizonans are diabetic or pre-diabetic resulting in $6.4 billion in health care and productivity costs. The severity and incidence of Type 2 Diabetes Mellitus (T2DM) is directly related to the hepatic lipid concentration. The degree of hepatic lipid accumulation is communicated by the hepatic vagal afferent nerve (HVAN) to regulate pancreatic insulin secretion and whole body insulin sensitivity. We have shown that obesity enhances expression of GABA-Transaminase (GABA-T) decreasing hepatic release of the excitatory neurotransmitter, aspartate, and increasing release of the inhibitor neurotransmitter, GABA. This enhanced inhibitory tone decreases hepatic vagal afferent nerve activity, increasing pancreatic insulin release and decreasing skeletal muscle glucose clearance/insulin sensitivity. Pharmacological inhibition of GABA-T robustly improves glucose homeostasis in diet induced obese mice. We propose 2 clinical objectives that will test the effect of GABA-T inhibition on glucose tolerance and insulin sensitivity in obese, hyperglycemic, hyperinsulinemic patients.

DETAILED DESCRIPTION:
Experimental Design: Hyperglycemic, hyperinsulinemic and mildly hypertensive (taking medication for hypertension or with systolic blood pressure of ≥135 mmHG) adult patients (18-60 y) with BMI ≥ 25 on insulin or metformin only and will be recruited using existing relationships between community partners and the University of Arizona Division of Endocrinology. Patients will be stratified into 2 treatments (Vigabatrin or Placebo) based on age, sex, and HbA1c (day -24).

For each treatment, Vigabatrin and placebo participants will be stratified as such: Each group will have equal distribution of male and female participants and each group will have similar HbA1c. This is a double-blind study and only the research pharmacist and Dr. Renquist will know which participants receive Vigabatrin or Placebo treatments. Dr. Renquist will be the one to place subjects into each treatment group using the guideline mentioned above.

Study Visit 1: (day -24; relative to treatment initiation) Dr. Herbst will be present to discontinue metformin and initiate a monitoring plan. Participants on long acting insulin will stop taking insulin 3 days prior to visits 2,3,4 and 5 and those on short acting insulin with stop taking insulin 12 hours prior to visits 2,3,4 and 5. On day (-24), patients will enter the CaTS (Clinical and Translational Science) Center after an overnight fast without having taken the blood pressure medication (if on any) that morning for a baseline assessment of body weight, height and blood pressure along with temperature, heart rate, O2 and respiration. A fasting blood sample will be collected into EDTA tubes to allow for measurement of plasma insulin, c-peptide, glucose, glucagon, and GABA. Following centrifugation (15 min, 3000xg) plasma will be aliquoted into 10 individual samples that will be immediately frozen at -80C for analyses in the Renquist laboratory. A peripheral vision field test will be performed on all participants and urine pregnancy test will be performed on female participants. A medical history will be taken from the subjects (self disclosure) and physical examination will be done. At this time, participants will be given a ledger in which to note daily blood glucose taken after an overnight fast for those on metformin. Participants taking insulin will note daily blood glucose taken after an overnight fast and immediately prior to lunch and dinner for the entire study (3 times daily). If fasting blood glucose rises more than 30 mg/dL after discontinuing metformin treatment (occurs in less than 5% of patients), patients will be advised to resume metformin treatment and visit their primary care physician. They will also be withdrawn from the study at this time. If it is after hours and they have concerns related to glucose levels, and are unable to reach clinical staff, they will be informed to go to the nearest Emergency Department, if they consider it to be an emergency. Participants will also be asked to not donate blood, change their physical activity habits or start a weight loss program while part of the study. This visit will take approximately 2 hours.

Study Visit 2: (Day -3 relative to treatment initiation) Three weeks after the initial visit (day -3 ), study participants will arrive at the CaTS Center after an overnight fast without having taken the blood pressure medication (if on any) that morning . They will have been reminded to stop taking insulin 3 days or 12 hours prior depending if they are on long acting insulin or short acting insulin, respectively. Time, temperature, heart rate, O2, respiration along with body weight, blood pressure, and a fasting blood sample will be collected (15 min after Peripheral IV insertion). Urine pregnancy test will also be done on female participants. The ledger will be examined to ensure that the participants are recording information appropriately and completely. We will subsequently perform the 2h, 7 sample glucose tolerance test (OGTT). Patients will be given a solution containing 75 g glucose to consume within 3 minutes. Blood samples will be collected at 0, 10, 20, 30, 60, 90, and 120 minutes for measurement of plasma glucose, insulin, and c-peptide. Once the glucose is back to 300mg/dl or lower, participants will be allowed to leave for the day. This visit will take approximately 3 hrs.

Study Visit 3: (day 0, relative to treatment initiation) 3 days post OGTT (day 0), participants will again arrive at the CaTS Center after an overnight fast without having taken the blood pressure medication (if on any) that morning. They will have been reminded to stop taking insulin 3 days or 12 hours prior depending if they are on long acting insulin or short acting insulin, respectively. Urine pregnancy test will also be done for female participants. Clinical lab personnel will take time, temperature, heart rate, O2, respiration along with body weight, blood pressure and collect fasting blood for measure of plasma insulin, glucose, glucagon, c-peptide and HbA1c (15 min after Peripheral IV insertion.) Participants' arm with IV will be place inside a heated box the entire study to promote blood flow. Subsequent to baseline measures, CaTS staff will perform hyperinsulinemic euglycemic clamps. Glucose tracer infusion will start and will be given continuously. 2 hours after the tracer infusion, Insulin will be intravenously infused at 80 mU/m2/min (dose per body surface area per minute). This infusion rate will result in a hyperinsulinemic state, simultaneously increasing glucose disposal into skeletal muscle and adipose tissue and depressing hepatic glucose production. Blood glucose is monitored every 5 minutes and 20% D-Glucose with a 6,6-2H2 Glucose tracer will be infused at a variable rate to maintain euglycemia. After at least 1 hour of constant insulin infusion, steady state conditions for plasma insulin, blood glucose and the glucose infusion rate will be achieved. Steady state will be defined as a glucose infusion rate that varies less than 5% for at least 30 minutes. Insulin and glucose infusion will be done for 2 hours once insulin infusion starts. At least 4 samples will be taken at 10 minute intervals during the steady state conditions for analysis of 2H-labeled glucose. Dilution of the 6,6-2H2 glucose relative to total glucose in the blood will indicate the rate of hepatic glucose production. The hepatic glucose production rate + glucose infusion rate sum to equal whole-body glucose clearance. Participants will be given lunch after study is finished. Subsequently, patients will be given either placebo or vigabatrin to be taken over the following weeks. Participants will be asked to come in at the end of each week to refill their medication and conduct a brief visit with nursing staff at CaTS. Patients will be instructed to take1 pill 2X/day for the first 7 days (days 0-6; 1000mg/day), 2 pills 2X/day for days 7-13 (2000mg/day), and three pills 2X/day for days 14-23 (3000mg/day). This visit will take approximately take 5 hours.

Brief visit 1, 2: (days 7 and 14, relative to treatment initiation) Medication will be refilled and dosage will be increased each week. Participants will speak to the nurses (Alma D-Leon, RN and Guadalupe E-Ortega, MSN, ACNP-BC) about general health and compliance with medication regiment.

Study Visit 4: (day 21, relative to treatment initiation) Participants will again arrive at the CaTS Center after an overnight fast without having taken the blood pressure medication (if on any) that morning. Time, temperature, heart rate, O2, respiration along with body weight, blood pressure, and a fasting blood sample will be collected. They will have stopped taking insulin 3 days or 12 hours prior depending if they are on long acting insulin or short acting insulin, respectively. A urine pregnancy test will also be done for female participants. The ledger will be examined to ensure that the participants are recording information appropriately and completely. The OGTT and all performed on day -3 (Study Visit 2) will be repeated on day 21. This visit will take approximately 3 hours.

Study Visit 5: (Day 24, relative to treatment initiation). Participants will again arrive at the CaTS Center after an overnight fast without having taken the blood pressure medication (if on any) that morning. They will have been reminded to stop taking insulin 3 days or 12 hours prior depending if they are on long acting insulin or short acting insulin, respectively. Their ledger will be reviewed. A peripheral vision field test will be performed on all participants. Temperature, heart rate, O2, respiration along with body weight, blood pressure, and a fasting blood sample will be collected (15 min after Peripheral IV insertion). The hyperinsulinemic-euglycemic clamp performed on day 0 (Study Visit 3) will be repeated on day 24. Beginning on day 24, participants on the vigabatrin and placebo treatment will initiate the step-down as recommended by the manufacturer, moving to the 2 pill 2X/day dose for days 24-30, and 1 pill 2X/day dose for days 31-37 before discontinuing treatment. Participants will be asked to come in at the end of each week to refill their medication and a brief visit with nursing staff at CaTS. Throughout the study, participants and lab personnel will be blinded to treatments. This visit will take approximately 5 hours.

Brief visit 3: (Day 31, relative to treatment initiation) Medication will be refilled and dosage will be decreased each week. Participants will speak to the nurses (Alma D-Leon, RN and Guadalupe E-Ortega, MSN, ACNP-BC) about general health and compliance with medication regiment.

Study Visit 6: (Day 45, relative to treatment initiation) On day 45, 1 week after the last dose of vigabatrin or placebo, patients on the vigabatrin and placebo treatment will be seen for an exit evaluation. Participants will again arrive at the CaTS Center after an overnight fast without having taken the blood pressure medication (if on any) that morning. Clinical lab personnel will take temperature, heart rate, O2, respiration, body weight and blood pressure and collect fasting blood for measure of plasma insulin, glucose, glucagon, c-peptide and HbA1c. A peripheral field vision test will be performed on all participants. The ledger of blood glucose measures will be collected for study analysis. Participants will be scheduled to follow up for vision exam within 6 months of study completion. This visit will take approximately 2 hours.

Timeline of proposed study, including Oral glucose tolerance tests (OGTT) and hyperinsulinemic euglycemic clamps (HEC). Weeks and days are numbered relative to treatment initiation.

Blood Samples Collected

Baseline samples:

Blood samples (< 10 mL) will be collected on days -24, -3, 0, 21, 24, and 45.

During oral glucose tolerance test:

Blood samples (< 10 mL) will be collected at 0, 10, 20, 30, 60, 90, and 120 minutes. Total blood < 100mLs.

During Hyperinsulinemic euglycemic clamps:

Blood samples (<10 mL) will be collected at times -120, -30, -20, -10, 0 and +90, +100, +110 and +120.

Risks

During the Informed Consent process, study personnel will address potential discomfort and risks associated with the study protocol. These will be included in the Informed Consent form.

ELIGIBILITY:
Inclusion Criteria:

* Participants that have BMI ≥ 25
* Participants that are mildly hypertensive(≥135 mm HG systolic BP) or taking medication for hypertension
* Hyperglycemic, hyperinsulinemic adults (18-60 y) on insulin or metformin only will be recruited based on elevated HbA1c using existing relationships between community partners and the University of Arizona Division of Endocrinology.
* Patients will be stratified into 2 treatments (Vigabatrin or Placebo) based on age, sex, and HbA1c taken at d -24.

Exclusion Criteria:

* BMI < 25
* Insulin Sensitive Individuals
* Participants with normal blood pressure (120/80 mm HG)
* Participants on any other diabetes therapy besides metformin and insulin
* If Pregnant or breast feeding
* If participants smoke
* Individuals who have complex partial seizures
* Individuals who are on other drugs to help with retinopathy or glaucoma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2030-04-15 (Estimated); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Fasted serum glucose and insulin | 3 weeks after treatment initiation
  Overnight fasted serum glucose and insulin
Glucose Clearance | 3 weeks after treatment initiation
  Clearance of glucose during an oral glucose tolerance test
Insulin Sensitivity | 24 days after treatment initiation
  Insulin sensitivity measured by glucose infusion rate required to maintain euglycemia during a hyperinsulinemic clamp
Blood Pressure | 21 days after treatment initiation
  Measure basal blood pressure both before and 21 days after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Renquist, PhD, Principal Investigator — University of Arizona

IPD SHARING:
Plan to Share IPD: No